CLINICAL TRIAL: NCT00493636
Title: A Double-Blind, Randomized Phase 2b Study of Sorafenib Compared to Placebo When Administered in Combination With Chemotherapy for Patients With Locally Advanced or MBC That Has Progressed During or After Bevacizumab Therapy
Brief Title: 1st or 2nd Line MBC (Metastatic Breast Cancer) With Previous Avastin (Bevacizumab) Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACORN AC01B07
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Sorafenib; Sugars; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Sorafenib + Gemcitabine or Capecitabine) (Active Comparator): Sorafenib will be administered (400 mg; 2 tablets x 200 mg) orally twice daily (approximately every 12 hours); Gemcitabine will be administered 1000 mg/m2 pm Days 1 and 8 of a 21 day cycle; Capecitabine will be administered orally at a dose of 1,000 mg/m2 twice daily, within 30 minutes after a meal, for 14 days followed by a 7 day rest period (without capecitabine)
  Interventions: Drug: Gemcitabine; Drug: Sorafenib; Drug: Capecitabine
- B (Placebo + Gemcitabine or Capecitabine) (Placebo Comparator): Placebo will be administered ( 2 tablets ) orally twice daily (approximately every 12 hours); Gemcitabine will be administered 1000 mg/m2 pm Days 1 and 8 of a 21 day cycle; Capecitabine will be administered orally at a dose of 1,000 mg/m2 twice daily, within 30 minutes after a meal, for 14 days followed by a 7 day rest period (without capecitabine)
  Interventions: Drug: Gemcitabine; Drug: Placebo; Drug: Capecitabine

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine will be administered 1000 mg/m2 pm Days 1 and 8 of a 21 day cycle
  Other Names: Gemzar
Drug: Sorafenib — Sorafenib will be administered (400 mg; 2 tablets x 200 mg) orally twice daily (approximately every 12 hours)
  Other Names: Nexavar
  Arms: A (Sorafenib + Gemcitabine or Capecitabine)
Drug: Placebo — Placebo will be administered (400 mg; 2 tablets x 200 mg) orally twice daily (approximately every 12 hours)
  Other Names: Sugar pill
  Arms: B (Placebo + Gemcitabine or Capecitabine)
Drug: Capecitabine — Capecitabine will be administered orally at a dose of 1,000 mg/m2 twice daily, within 30 minutes after a meal, for 14 days followed by a 7 day rest period (without capecitabine).
  Other Names: Xeloda

SUMMARY:
The study is being conducted to compare progression-free survival in patients treated with sorafenib and gemcitabine/capecitabine versus patients treated with placebo and gemcitabine/capecitabine for locally advanced or metastatic breast cancer that has progressed during or following treatment with a bevacizumab-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast.
* Measurable or evaluable locally advanced or metastatic disease.
* Age ≥18 years.
* Disease progression during or after treatment with a bevacizumab-containing regimen in the adjuvant or first-line metastatic setting.
* Patients must have discontinued chemotherapy at least 3 weeks prior to randomization.
* No more than one prior chemotherapy regimen for locally advanced or metastatic disease.
* Prior hormonal therapy allowed provided it has been discontinued prior to randomization.
* Prior radiation therapy is allowed but must be completed at least 3 weeks prior to randomization. Previously radiated area(s) must not be the only site of disease.
* ECOG Performance Status of 0 or 1.
* Adequate bone marrow, liver, and renal function
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to randomization, and must agree to use adequate contraception prior to study entry, for the duration of study participation and 28 days after the last study drug dosing.
* Patients must be able and willing to sign a written informed consent.
* Patients must be able to swallow and retain oral medication.

Exclusion Criteria:

* Patients with breast cancer over-expressing human epidermal growth factor receptor 2 (HER-2) (gene amplification by FISH or 3+ over-expression by immunohistochemistry). Patients with unknown HER-2 status are not eligible.
* Patients with active brain metastases.
* Major surgery, open biopsy, or significant traumatic injury within 4 weeks of randomization.
* Prior use of gemcitabine/capecitabine or sorafenib.
* Evidence or history of bleeding diathesis or coagulopathy.
* Serious, non-healing wound, ulcer, or bone fracture.
* Substance abuse, or medical, psychological, or social condition that may interfere with the patient's participation in the study or evaluation of the study results.
* Use of cytochrome P450 enzyme-inducing anti-epileptic drugs is not allowed.
* Clinically significant cardiac disease
* Uncontrolled hypertension
* Thrombolic, embolic, venous, or arterial events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event > NCI-CTCAE Grade 2 within 4 weeks of randomization.
* Any other hemorrhage/bleeding event ≥ NCI-CTCAE Grade 3 within 4 weeks of randomization.
* Active clinically serious infection > NCI-CTCAE Grade 2.
* Known HIV infection or chronic hepatitis B or C (the safety and effectiveness of sorafenib in this patient population have not been studied).
* Previous or concurrent cancer that is distinct in primary site or histology from breast cancer EXCEPT cervical cancer in-situ, treated basal cell carcinoma, superficial bladder tumors [Ta and Tis] or any cancer curatively treated > 5 years prior to randomization.
* Known or suspected allergy to sorafenib or gemcitabine/capecitabine.
* Prior or concurrent use of St. John's Wort or rifampin (rifampicin) within 3 weeks of randomization.
* Concurrent anti-cancer therapy other than gemcitabine/capecitabine and sorafenib/placebo.
* Prior treatment with any agent that targets VEGF or VEGFR (licensed or investigational), except bevacizumab.
* Women who are pregnant or breast-feeding.
* Use of any investigational drug within 30 days or 5 half-lives, whichever is longer, preceding randomization.
* Inability to comply with protocol and/or not willing or not available for follow-up assessments.
* Any condition which in the investigator's opinion makes the patient unsuitable for the study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-06; Primary Completion 2010-09 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Schwartzberg, MD, FACP, Study Chair — Accelerated Community Oncology Research Network Inc; Clifford A Hudis, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (44):
- United States (44):
  - Providence Cancer Center / Katmai Oncology Group LLC, Anchorage, Alaska
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Compassionate Cancer Care-Corona, Corona, California
  - Compassionate Cancer Care-Fountain Valley, Fountain Valley, California
  - California Cancer Care, Greenbrae, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Compassionate Cancer Care-Riverside, Riverside, California
  - Sutter Cancer Center, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco Comprehensive Cancer Center, San Francisco, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Hematology Oncology PC / Bennett Cancer Center, Stamford, Connecticut
  - Oncology Associates of Bridgeport, Trumbull, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Pasco Hernando Oncology Associates PA, Brooksville, Florida
  - Pasco Hernando Oncology Associates PA, New Port Richey, Florida
  - Augusta Oncology Associates, PC, Augusta, Georgia
  - Cascade Cancer Center, Macon, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Northwest Georgia Oncology Center, Marietta, Georgia
  - Northwestern University-Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Columbia Comprehensive Cancer Care Clinic & Research Institute, Jefferson City, Missouri
  - Oncology Hematology Specialists, PA, Denville, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of New York, East Syracuse, New York
  - Queens Cancer Center, Jamaica, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - North Coast Cancer Care, Sandusky, Ohio
  - Hematology Oncology of Northeast Pennsylvania, Dunmore, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - The West Clinic, Memphis, Tennessee
  - Oncology Alliance, Glendale, Wisconsin

REFERENCES:
- [Derived] Schwartzberg LS, Tauer KW, Hermann RC, Makari-Judson G, Isaacs C, Beck JT, Kaklamani V, Stepanski EJ, Rugo HS, Wang W, Bell-McGuinn K, Kirshner JJ, Eisenberg P, Emanuelson R, Keaton M, Levine E, Medgyesy DC, Qamar R, Starr A, Ro SK, Lokker NA, Hudis CA. Sorafenib or placebo with either gemcitabine or capecitabine in patients with HER-2-negative advanced breast cancer that progressed during or after bevacizumab. Clin Cancer Res. 2013 May 15;19(10):2745-54. doi: 10.1158/1078-0432.CCR-12-3177. Epub 2013 Feb 26. PMID 23444220

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The period of study was 28 Jun 2007 (first subject randomized) to 29 Feb 2012 (overall survival data cutoff date). There were 40 centers in the United States that participated in this trial.
Pre-assignment Details: 181 patients were assessed for eligiblity. Of these, 21 patients were excluded from the trial due to not meeting the eligibility criteria, leaving 160 patients who were randomized.
Period: Overall Study
Arm/Group | A (Sorafenib + Gemcitabine or Capecitabine) | B (Placebo + Gemcitabine or Capecitabine)
Started | 81 | 79
Completed | 79 | 77
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease progression/recurrence/relapse | 0 | 1
Not completed — Mis-randomization | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients are included (i.e., the intent-to-treat population)
Groups:
- Total: Total of all reporting groups
Arm/Group | A (Sorafenib + Gemcitabine or Capecitabine) | B (Placebo + Gemcitabine or Capecitabine) | Total
Number analyzed (Participants) | 81 | 79 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (10.6) | 54.2 (11.0) | 53.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 79 | 160
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 81 | 79 | 160

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Time Frame: From the date of randomization to date of first documented disease progression (i.e., the date on which a radiologic procedure or clinical evaluation was performed) or the date of death due to any cause, if before progression, assessed up to 39 months.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | A (Sorafenib + Gemcitabine or Capecitabine) | B (Placebo + Gemcitabine or Capecitabine)
Number analyzed (Participants) | 81 | 79
Days | 103 [83 to 128] | 81 [48 to 95]

2. Secondary Outcome: Overall Survival
Time Frame: From the date of randomization to date of death due to any cause, assessed up to 56 months.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | A (Sorafenib + Gemcitabine or Capecitabine) | B (Placebo + Gemcitabine or Capecitabine)
Number analyzed (Participants) | 81 | 79
Days | 407 [308 to 492] | 348 [297 to 457]

3. Secondary Outcome: Time to Progression
Time Frame: Calculated as the time (days) from date of randomization to date of first observed disease progression (radiological or clinical, whichever is earlier), assessed up to 39 months.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | A (Sorafenib + Gemcitabine or Capecitabine) | B (Placebo + Gemcitabine or Capecitabine)
Number analyzed (Participants) | 81 | 79
Days | 111 [85 to 128] | 82 [48 to 95]

4. Secondary Outcome: Overall Response Rate
Description: Overall response rate was defined as the proportion of participants experiencing complete response (CR) and partial response (PR) as best overall response. Response was evaluated via changes from baseline in radiological tumor measurements using RECIST version 1.0 guidelines, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter (LD) of target lesions; Stable Disease (SD) is neither sufficient shrinkage in sum of LD of target lesions to be PR nor increase of >=20%; Progressive Disease (PD) is the increase in existing lesions or new lesions.
Time Frame: The overall tumor burden at baseline will be compared with subsequent measurements up to the date of first documented disease progression or the date of death due to any cause, if before progression, assessed up to 39 months.
Measure: Number; unit: percentage of participants
Arm/Group | A (Sorafenib + Gemcitabine or Capecitabine) | B (Placebo + Gemcitabine or Capecitabine)
Number analyzed (Participants) | 81 | 79
percentage of participants | 19.8 | 12.7

5. Secondary Outcome: Duration of Overall Response
Description: Duration of overall response was calculated as the time (days) from first documentation of CR or PR (whichever status is recorded first) until the first date that recurrent or progressive disease (PD) or death is objectively documented. Response was evaluated via changes from baseline in radiological tumor measurements using RECIST version 1.0 guidelines, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter (LD) of target lesions; Stable Disease (SD) is neither sufficient shrinkage in sum of LD of target lesions to be PR nor increase of >=20%; Progressive Disease (PD) is the increase in existing lesions or new lesions.
Time Frame: Period measured from the first documentation of complete or partial response (whichever status is recorded first) until the first date that recurrent or progressive disease or death is objectively documented.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | A (Sorafenib + Gemcitabine or Capecitabine) | B (Placebo + Gemcitabine or Capecitabine)
Number analyzed (Participants) | 81 | 79
Days | 94 [68 to 134] | 147 [86 to 372]

ADVERSE EVENTS:
Arm/Group | A (Sorafenib + Gemcitabine or Capecitabine) | B (Placebo + Gemcitabine or Capecitabine)
Serious Adverse Events (participants affected / at risk) | 32/79 | 28/77
Other Adverse Events (participants affected / at risk) | 78/79 | 73/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A (Sorafenib + Gemcitabine or Capecitabine) (N=79) | B (Placebo + Gemcitabine or Capecitabine) (N=77)
Vomiting (Gastrointestinal disorders) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 5
Cellulitis (Infections and infestations) | 0 | 2
Disease progression (General disorders) | 2 | 2
Pyrexia (General disorders) | 1 | 3
Fatigue (General disorders) | 3 | 0
Mucosal inflammation (General disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A (Sorafenib + Gemcitabine or Capecitabine) (N=79) | B (Placebo + Gemcitabine or Capecitabine) (N=77)
Nausea (Gastrointestinal disorders) | 35 | 38
Diarrhea (Gastrointestinal disorders) | 29 | 17
Constipation (Gastrointestinal disorders) | 18 | 21
Vomiting (Gastrointestinal disorders) | 21 | 18
Stomatitis (Gastrointestinal disorders) | 21 | 5
Abdominal pain (Gastrointestinal disorders) | 11 | 10
Abdominal distension (Gastrointestinal disorders) | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Fatigue (General disorders) | 49 | 38
Pyrexia (General disorders) | 15 | 16
Pain (General disorders) | 11 | 8
Mucosal inflammation (General disorders) | 11 | 5
Edema peripheral (General disorders) | 7 | 5
Chest pain (General disorders) | 6 | 5
Chills (General disorders) | 5 | 4
Asthenia (General disorders) | 2 | 5
Influenza like illness (General disorders) | 4 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 45 | 14
Rash (Skin and subcutaneous tissue disorders) | 22 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Headache (Nervous system disorders) | 19 | 14
Dizziness (Nervous system disorders) | 5 | 10
Neuropathy (Nervous system disorders) | 6 | 2
Dysgeusia (Nervous system disorders) | 5 | 1
Neuropathy peripheral (Nervous system disorders) | 4 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 5
Paresthesia (Nervous system disorders) | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 19 | 21
Anemia (Blood and lymphatic system disorders) | 12 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 8
Leukopenia (Blood and lymphatic system disorders) | 5 | 5
Weight decreased (Investigations) | 11 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 7
Alanine aminotransferase increased (Investigations) | 5 | 5
Neutrophil count decreased (Investigations) | 5 | 3
Hemoglobin abnormal (Investigations) | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 15 | 7
Dehydration (Metabolism and nutrition disorders) | 7 | 4
Hypokalemia (Metabolism and nutrition disorders) | 5 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 4
Pneumonia (Infections and infestations) | 2 | 6
Sinusitis (Infections and infestations) | 4 | 2
Hypertension (Vascular disorders) | 16 | 7
Hot flush (Vascular disorders) | 6 | 3
Deep vein thrombosis (Vascular disorders) | 5 | 1
Anxiety (Psychiatric disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Onyx has the right to require the deletion of any "Confidential Information" in a publication. If Onyx believes that information contained in the publication is patentable and communicates that in writing, the submission/delivery of the publication may be delayed for up to 60 additional days to allow for the filing of a United States (and any other appropriate) patent application(s).